CLINICAL TRIAL: NCT05440721
Title: Clinical Trial of an Innovative Digital Therapeutic for Smoking Cessation With Biochemical Verification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of company's priority; learning from a separate CT-101-CLS-001 (NCT04857515) is deemed sufficient
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CT-101-002
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Nicotine Addiction; Drug Addiction; Drug Dependence; Substance Use Disorder; Tobacco Dependence
Keywords: Smoking; Cigarette Smoking; Tobacco Smoking; Nicotine; Drug; Addiction; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Smoking; Cigarette Smoking; Tobacco Smoking; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment A (device Clickotine®) (Active Comparator): User will open and use Treatment A (Clickotine® device) several times a day up to their quit date to complete a program of 21 Missions.
  Interventions: Device: Treatment A with device Clickotine® (Active intervention)
- Treatment B (smoking education) (Sham Comparator): Treatment B app provides education and support to smokers seeking to quit. When a user has a craving or wants support or education, they can log into the app.
  Interventions: Device: Treatment B with smoking education (control)

INTERVENTIONS:
Device: Treatment A with device Clickotine® (Active intervention) — The intervention regimen around Treatment A is almost entirely user-directed. When a person has a craving, a series of options are available to ease the craving and resist the urge to smoke. The user will also engage with Clickotine® leading up to their quit date to complete a program of 21 Missions, daily activities which help prepare them to quit and keep them off cigarettes. Ideally, the user will open and use Treatment A several times a day.
  Arms: Treatment A (device Clickotine®)
Device: Treatment B with smoking education (control) — The Treatment B app is operated by the National Cancer Institute to provide education and support to smokers seeking to quit. The QG regimen is entirely user-directed. When a user has a craving or wants support or education, they can log into the QG app. The QG app also provides lessons relevant for preparing to quit and beginning to quit.
  Arms: Treatment B (smoking education)

SUMMARY:
This study is evaluating the efficacy of Treatment A for short-term smoking cessation through a blinded randomized controlled trial (RCT) vs.Treatment B.

DETAILED DESCRIPTION:
The overarching study aim is to recruit a population of current smokers who are motivated to quit with the assistance of a mobile solution, enroll them into a study testing apps to help them quit, and randomize them into one of two arms. The core study period will consist of 8 weeks of usage of Treatment A or Treatment B. At the end of this period, users will receive notifications to link them to an online survey, which will record their responses in a secure database.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65
2. Smokes at least 5 cigarettes daily
3. Is interested in quitting in the next 30 days
4. Owns an iPhone with iOS 9 or higher or Android with OS 4.1 or higher
5. Willing and able to receive SMS text messages
6. Able to comprehend the English-language and the informed consent form
7. Lives in the United States
8. One half of the study sample will be recruited from the general population of smokers via social media advertisements
9. One half of the study sample will be recruited via mail from a Magellan Behavioral Health value-based care network

Exclusion Criteria:

1. Prior use of Clickotine or QuitGuide
2. Current use of pharmacotherapy for smoking cessation or nicotine replacement therapy (NRT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: | [Time Frame: 8 week core study]
  The primary objective is to confirm the improved efficacy of CKT for short-term smoking cessation through a blinded randomized controlled trial (RCT) vs. QuitGuide.
  **Acceptance criteria: Self-reported 30 day point prevalence quit rates will be significantly higher in the CKT arm than QuitGuide.

SECONDARY OUTCOMES:
Secondary Outcome Measure | [Time Frame: 8 week core study]
  A secondary objective of the study is to establish the feasibility of biochemical verification of smoking cessation in a fully remote, digital clinical trial.
Secondary Outcome Measure | [Time Frame: 8 week core study]
  A secondary objective of the study is to compare cessation rates between the CKT+NRT group and the CKT-only group, to address expected med/NRT use during the trial and to confirm the initial trial result that CKT+NRT is not superior to CKT-alone.
Secondary Outcome Measure | [Time Frame: 8 week core study]
  A secondary objective of the study is to demonstrate the feasibility of evaluating CKT in a Magellan Behavioral Health (A Click Therapeutics partner) value-based care population

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MDPhD, FAAN, Study Chair — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No